CLINICAL TRIAL: NCT05199987
Title: Impact of Occupational Therapy With Breathing Control Exercises in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Breathing Control Exercises in Patients With Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ErgoControl
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Severe Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Occupational therapy; Breathing control
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Occupational Therapy (Active Comparator): This group will receive standard occupational therapy sessions
  Interventions: Behavioral: Standard Occupational Therapy
- Occupational Therapy with Breathing Control Exercises (Experimental): This group will receive the same component of the control group + breathing control exercises
  Interventions: Behavioral: Occupational Therapy with Breathing Control Exercises

INTERVENTIONS:
Behavioral: Standard Occupational Therapy — Standard occupational therapy sessions include patient therapeutic education (implementation of strategies and/or technical aids promoting autonomy and independence), walking and stair exercises in real-life conditions (weighted shopping bag, unstable ground, ...), as well as work on activities of daily living aiming to improve toileting skills (includes individual assessment, the use of technical aids depending of this assessment, and personalised strategies to conserve energy).
  Arms: Standard Occupational Therapy
Behavioral: Occupational Therapy with Breathing Control Exercises — Includes the same treatment than the one described in standard occupation therapy but with the addition of 30-minute sessions per day on breathing control exercises. These exercises included the reproduction of gestures reproducing daily activities and simultaneous explanations of breathing techniques that the patient can perform in order to set up strategies for saving breath during exercise.
  Arms: Occupational Therapy with Breathing Control Exercises

SUMMARY:
The purpose of this study is to test whether breathing control exercises embedded in occupational therapy sessions have an impact on quality of life and dyspnea in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Dyspnea is one of the most important and debilitating symptoms in patients with COPD and is often the starting point to the vicious cycle of physical inactivity. As a consequence of increased dyspnea, patients adapt themselves by reducing the amount of all activities of daily living performed, with a consequent reduction in quality of life.

Occupational therapists are involved in pulmonary rehabilitation programs aiming to improve the biopsychosocial condition of COPD patients. However, the specific roles and intervention of occupational therapists are not well-defined, and standardized protocols are lacking. The implementation of breathing control exercises in occupational therapy sessions, aiming among other things to regulate patient's breathing during their activities of daily living, could be a starting point for a more effective management of patients with COPD. This could ultimately participate in the improvement of quality of life in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnostic of COPD
* Severity of COPD: global initiative for chronic obstructive lung disease (GOLD) classification III or IV
* Undergoing a pulmonary rehabilitation program in J. Bracops Hospital

Exclusion Criteria:

* Cardiac or orthopedic complications limiting participation in occupational therapy sessions
* Active smoking
* Inability to understand the French language orally or in writing
* Cognitive impairments limiting understanding of instructions and participation in occupational therapy sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change in St George's Respiratory Questionnaire score | At baseline and after 6 weeks of pulmonary rehabilitation
  Overall health, daily life, and perceived well-being are assessed via the St George's Respiratory Questionnaire and its three domains: "symptoms", "activities" and "impact".
  The score for each domain and the total score ranged from 0 to 100, with 100 indicating a very poor quality of life.

SECONDARY OUTCOMES:
Change in health-related quality of life | At baseline and after 6 weeks of pulmonary rehabilitation
  Health-related quality of life is assessed via the CAT (COPD assessment test) score. The assessment consists of eight questions, with a score associated with each question ranging from 0 to 5, with 0 indicating no impact on quality of life. The total score ranges from 0 to 40. The higher the score, the greater the impact on quality of life.
Change in dyspnea | At rest and after the effort, at baseline as well as after 6 weeks of pulmonary rehabilitation
  Dyspnea is rated with a visual analogic scale (0 to 100mm).
Change in hand grip strength | At baseline and after 6 weeks of pulmonary rehabilitation
  Hand grip strength test is assessed via a hand dynamometer (JAMAR). The best value of three repetitions of the best hand is reported.
Change in functional capacity | At baseline and after 6 weeks of pulmonary rehabilitation
  Functional capacity is assessed with the five-time sit-to-stand test. The time the individual takes to sit down and stand up completely over five repetitions is reported

CONTACTS AND LOCATIONS:
Locations (1):
- J Bracops Hospital, Anderlecht, Belgium